CLINICAL TRIAL: NCT04960384
Title: Fibroblast Growth Factor Regeneration of Tympanic Membrane Perforations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-00672
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — Fibroblast Growth Factor 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigator and the subject will be blinded to treatment assignment during the Randomized Treatment phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Human Fibroblast Growth Factor-2 (FGF-2) (Experimental)
  Interventions: Drug: FGF-2

INTERVENTIONS:
Drug: FGF-2 — The FGF-2 method of use comprises a pledget of gelatin sponge, with human fibroblast growth factor-2 (FGF-2) added to the pledget just before topical application to the tympanic membrane, and the use of fibrin glue used for applications in ear surgery. The concentration of the FGF-2 solution will be 100μg of FGF-2 per 1 mL with an estimated dose of about 20 μg in 0.2ml. Fibrin glue will be applied to secure gelatin sponge after placement according to the size of the membrane perforation. Application of the study treatment will occur at Visit 1 and may be repeated at each follow up visit as needed for a maximum of three treatments in the Randomized Treatment Phase (Visit 1, Visit 2, and Visit 3).
  Arms: Human Fibroblast Growth Factor-2 (FGF-2)
Drug: Placebo — FGF-2 will be replaced with sterile water to saturate a pledget of gelatin sponge. The method will be otherwise identical to the FGF-2 intervention.
  Arms: Placebo

SUMMARY:
This study is a double blinded, placebo-controlled phase II study evaluating the efficacy of FGF-2 for the treatment of chronic non-healing tympanic membrane perforations (TMP). The documentation of TM closure will be the main efficacy outcome measure. Pretreatment photographs will document the area of the TM perforation and allow measurement of surface areas of the TMP for comparison of pre- and post-treatment. The study will be divided into two phases, the Randomized Treatment phase (part A), and the Unblinded Crossover phase (part B). In part A of the study, subjects will be randomized 1:1 (using simple randomization) to receive FGF-2 or placebo treatment up to 3 treatments. Subjects that fail three study treatments will move on to part B of the study. Subjects who received placebo in part A and failed three placebo treatments will crossover to receive unblinded FGF-2 for up to 3 treatments. Subjects who received FGF-2 in part A and failed three experimental treatments will not have additional FGF-2 treatment, and will move on to study follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Dry tympanic membrane perforation of at least 6 months duration
* Any person of child-bearing potential, must have a negative beta-HCG test and must agree to use an adequate form of birth control throughout the clinical trial.

Exclusion Criteria:

* Active otitis media or chronic otorrhea from the middle ear
* Subjects receiving radiation therapy, corticosteroids, immunosuppressive agents, or chemotherapy
* Subjects who, at study entry, are taking systemic antibiotics
* Subjects who are immunosuppressed
* Subjects experiencing bacterial or viral infection or who may otherwise be febrile or may be with inflammation.
* Life expectancy of less than 1 year
* Active alcohol or drug abuse within 6 months prior to study entry
* Significant medical condition that could prevent full participation in the procedures required for the study
* Known or suspected allergies to any components used in the study, i.e. porcine collagen
* Subjects who have cholesteatoma mass, or endothelium invasion in the tympanic cavity
* Subjects whose total perforation cannot be seen by an endoscope
* Subjects with inadequately controlled diabetes mellitus (NGSP: HbA1c 6.9% or higher)
* Subjects with a history of malignant ear canal tumors within 3 years of screening for eligibility
* Subjects who have undergone prior myringoplasty or tympanoplasty
* Subjects whose TMP is a result of thermal burn, or radiation therapy.
* Subjects who have abnormalities in the auditory ossicles or their linkages
* Subjects having moderate to severe dementia such as Alzheimer's disease or senile dementia
* Subjects whose hearing ability does not improve to bone-conduction hearing on a hearing acuity test using the tentative closure of perforation with a wet cotton ball.
* Subject having residual TM with abnormal form or abnormal shape anatomically
* Subjects having any granulation or soft tissue density due to inflammation, or infection in mastoid antrum determined by CT scanning (Temporal bone CT scanning)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
TMP Closure Ratio | up to Day 134
  Determined by otoscopic exam and photographic documentation

SECONDARY OUTCOMES:
Time to Closure of TMP | up to Day 134
Pure-tone and speech discrimination scores | Pre-treatment (Day 1)
  Measured by audiograms (total range of score: 125, 250, 500, 1000, 2000, 4000, 8000 Hz). S
Pure-tone and speech discrimination scores | Post-treatment 1 (Day 22)
  Measured by audiograms (total range of score: 125, 250, 500, 1000, 2000, 4000, 8000 Hz). S
Pure-tone and speech discrimination scores | Post-treatment 1 (Day 43)
  Measured by audiograms (total range of score: 125, 250, 500, 1000, 2000, 4000, 8000 Hz). S
Pure-tone and speech discrimination scores | Post-treatment 1 (Day 64)
  Measured by audiograms (total range of score: 125, 250, 500, 1000, 2000, 4000, 8000 Hz). S
Pure-tone and speech discrimination scores | Post-treatment 1 (Day 85)
  Measured by audiograms (total range of score: 125, 250, 500, 1000, 2000, 4000, 8000 Hz). S
Pure-tone and speech discrimination scores | Post-treatment 1 (Day 106)
  Measured by audiograms (total range of score: 125, 250, 500, 1000, 2000, 4000, 8000 Hz). S
Pure-tone and speech discrimination scores | Post-treatment 1 (Day 127)
  Measured by audiograms (total range of score: 125, 250, 500, 1000, 2000, 4000, 8000 Hz). S
Pure-tone and speech discrimination scores | Post-treatment 1 (Day 134)
  Measured by audiograms (total range of score: 125, 250, 500, 1000, 2000, 4000, 8000 Hz). S
Air-Bone Gap (ABG) | up to Day 134
  Defined as the difference between air-conduction and bone-conduction audiometric thresholds
Mobility of the Tympanic Membrane | Day 134
  As measured by tympanometry
Salvage Rate of FGF-2 in Patients who Fail Placebo | Day 64

CONTACTS AND LOCATIONS:
Overall Officials: David Friedmann, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Only aggregate data will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to David.friedmann@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.